CLINICAL TRIAL: NCT04563013
Title: Study of the Effects of Transcutaneous Vagus Nerve Stimulation on Cancer Patients' Fatigue, Quality of Life and Lymphopenia After Radiotherapy or Chemotherapy
Brief Title: Study of the Effects of Transcutaneous Vagus Nerve Stimulation on Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xidian University (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Wei Qin, Professor, Xidian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20200110
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Cancer, Therapy-Related; Cancer-related Fatigue; Quality of Life
Keywords: Cancer-related fatigue; Transcutaneous vagus nerve stimulation; Breast cancer; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham taVNS (Sham Comparator): The participants under conventional radiotherapy were applied with sham taVNS at the left tragus with the power off for 30min. The intervention would last until to the end of conventional radiotherapy.
  Interventions: Device: Transcutaneous vagus nerve stimulation
- taVNS (Active Comparator): For taVNS group, the electrodes were attached to the tragus of left ear after skin preparation with an alcohol pad. The stimulation current was a single-phase rectangular pulse with the following stimulation parameters: duty circle: 60 s "on" periods and 10 s "off" periods; frequency: 30 Hz; pulse width: 200 μs; pulse amplitude of 0.5 mA to 1.5 mA; stimulation time:30 min.
  Interventions: Device: Transcutaneous vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation — the transcutaneous vagus nerve stimulation was conducted by ear clip with cathode and anode placed at the tragus for 30 min.

SUMMARY:
Patients diagnosed with breast cancer who received assisted radiotherapy were recruited and the transcutaneous auricular vagus nerve stimulation (taVNS) was applied. The aim of of study is : 1) to study whether taVNS could improve the patient's fatigue, quality of life under radiotherapy or chemotherapy; 2) to investigate the effects of taVNS on the levels of patients' lymphocyte subsets and proinflammatory cytokines.

DETAILED DESCRIPTION:
A prospective, randomized, double-blind, parallel controlled trial was conducted. This trail is to recruit 261 patients. Patients were randomly assigned in 2:1 ratio to two groups: 1) taVNS with conventional radiotherapy(intervention group); 2)sham taVNS with conventional radiotherapy (control group). taVNS was conducted at every radiotherapy day. taVNS stimulation method: for taVNS group, the electrodes were attached to the tragus of left ear after skin preparation with an alcohol pad, the stimulation current was a single-phase rectangular pulse with the following stimulation parameters: duty circle: 60 s "on" periods and 10 s "off" periods; frequency: 30 Hz; pulse width: 200 μs; pulse amplitude of 0.5 mA to 1.5 mA; stimulation time:30 min. For staVNS group, the clip electrodes were also placed on the left tragus but with no current output. The Fatigue Scale (BFI), the European Organization for Reasearch and Treatment of Cancer Quality of Life Questionnaire(EORTC QLQ-C30), Pittsburgh sleep quality index (PSQI) and Hospital Anxiety and Depression Scale (HADS) assessment, lymphocyte subpopulations,level of proinflammatory factors, blood routine testing and electrocardiogram testing were performed within 2 weeks before treatment (baseline), 4 weeks after intervention, end of chemoradiation and 1 month after the end of chemoradiation; weekly blood routine testing during intervention under radiotherapy and chemotherapy; the incidence of side effects and sleep quality score were evaluated at baseline, 2 weeks and 4 weeks after the intervention, at the end of radiotherapy and chemotherapy, and 1 month after the end of radiotherapy. The number of recruited participants met the statistical requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed with breast cancer, suitable for adjuvant radiotherapy after surgery;
2. Eastern Cooperative Oncology Group (ECOG) physical condition score: 0~1 point.

Exclusion Criteria:

1. Participants with organic brain lesions (cerebral hemorrhage, large-area cerebral infarction, encephalitis, epilepsy, etc.);
2. Participants with peptic ulcer, arrhythmia, or cardiac corrected QT interval> 450ms;
3. Participants who have slow breathing (less than 10 breaths per minute);
4. Participants who are or have been diagnosed with other major diseases (coronary heart disease, pulmonary heart disease, etc.);
5. Participants who are currently or have been diagnosed with mental disorders other than major depressive disorder;
6. Participants who are or have participated in vagus nerve or transcranial electrical stimulation treatment for less than 3 months;
7. Participants who are not suitable for vagus nerve stimulation treatment;
8. Participants who refuse to sign informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
the score of fatigue at 1 month | The taVNS treatment lasted about five weeks, data were collected at 1 month after the end of the taVNS treatment
  For fatigue degree evaluation, the Brief Fatigue Inventory (BFI) was used. The score of fatigue in two groups will be evaluated by BFI and will be compared. The scale uses the 11-point scoring method, whereby 0 points indicates no fatigue and 10 points the most severe fatigue. A higher score indicates more severe fatigue. The BFI included three fatigue severity items and six fatigue interference items. Three fatigue severity items ask patients to rate the severity of their fatigue at its "worst", "usual" and "now" during the past 24 h and another six fatigue interference items describe how much fatigue has interfered with different aspects of the patient's life during past 24 h, including general activity, mood, walking ability, normal work, relationships with other people and enjoy of life.

SECONDARY OUTCOMES:
the scores of HADS at End and at 1 month | The taVNS treatment lasted about five weeks, data were collected at the end of RT and taVNS treatment and 1 month after the end of taVNS treatment
  For depression and anxiety degree evaluation, the Hospital Anxiety and Depression Scale (HADS) was used. The HADS is a brief 14-item scale, with seven items in each of the anxiety and depression dimension scored from 0 to 3, resulting in scale scores ranging from 0 to 21.
the scores of PSQI at End and at 1 month | The taVNS treatment lasted about five weeks, data were collected at the end of RT and taVNS treatment and 1 month after the end of taVNS treatment
  For sleep evaluation, the Pittsburgh Sleep Quality Index (PSQI) was used. The PSQI was a 19-item self-report instrument that includes seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction.
the scores of EORTC QLQ-C30 at End and at 1 month | The taVNS treatment lasted about five weeks, data were collected at the end of RT and taVNS treatment and 1 month after the end of taVNS treatment
  The quality of life was evaluated by European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). It included a total of 30 entries, which were divided into 15 domains; among these, there were 5 functional domains (body, role, cognition, mood, and social function), 3 symptom domains (fatigue, pain, and nausea and vomiting), 1 overall health status/quality of life area and 6 single entries (each as a domain). The higher the score for the functional domains and overall health status, the better the functional status and quality of life. The final standardized score ranges from 0 to 100, with higher scores indicating better quality of life.
the change of cell counts of blood cells from baseline to End and to 1M. | The taVNS treatment lasted about five weeks, data were collected at the end of RT and taVNS treatment and 1 month after the end of taVNS treatment
  Clinical and laboratory parameters, including the cell counts of white blood cell, lymphocyte, neutrophil, platelet, the value of hemoglobin, were extracted from the electronic medical record for all patients.
the change in IL-6 level from baseline to End and to 1M. | The taVNS treatment lasted about five weeks, data were collected at the end of RT and taVNS treatment and 1 month after the end of taVNS treatment
  The levels of interleukin-6 (IL-6) was extracted from the electronic medical record for all patients.
the change in CRP level from baseline to End and to 1M. | The intervention lasted about five weeks, data were collected at the end of RT and taVNS treatment (End) and 1 month after the end of taVNS treatment (1M)
  The levels of C-reactive protein (CRP) was extracted from the electronic medical record for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Na Zhao, Doctor, Principal Investigator — the First Affiliated Hospital of the Air Force Medical University; Wei Qin, Doctor, Principal Investigator — Xidian University
Locations (1):
- Xidian University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
the data will be available by the publication of articles
Supporting Information: Study Protocol, CSR
Time Frame: The information will be available by the publication of articles